CLINICAL TRIAL: NCT00446979
Title: Phase I Study of the Safety and Acceptability of UC-781 Topical Vaginal Microbicide in Women and Acceptability in Their Male Partners,Chiang Rai, Thailand
Brief Title: Safety Study of UC-781 Vaginal Microbicide
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Centers for Disease Control and Prevention (U.S. Federal Agency)
Collaborators: Ministry of Health, Thailand (Other Government); CONRAD (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CDC-NCHHSTP-4744; MOPH 109/2548
Record Dates: First submitted 2007-03-12; First posted 2007-03-13 (Estimated); Last update posted 2013-04-19 (Estimated); Status verified 2013-04

CONDITIONS: HIV Infections
Keywords: Microbicides; HIV seronegativity
MeSH Terms: conditions — HIV Infections | interventions — UC-781

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): UC 781 0.1% carbomer gel
  Interventions: Drug: UC 781
- 2 (Experimental): UC 781 0.25% carbomer gel
  Interventions: Drug: UC 781
- 3 (Placebo Comparator): Placebo vaginal gel
  Interventions: Drug: Placebo gel

INTERVENTIONS:
Drug: Placebo gel — HEC (hydroxyethyl cellulose) Control Gel applied vaginally twice daily for two weeks
  Arms: 3
Drug: UC 781 — UC 781 0.1% or UC 781 0.25%, applied vaginally twice daily for two intermenstrual weeks
  Arms: 1; 2

SUMMARY:
This study will help determine whether UC-781 gel is safe when applied to the vagina twice daily for 14 days, and will assess whether women and men find the gel acceptable to use.

ELIGIBILITY:
Inclusion Criteria for women:

* Age 18-50 years old
* Regular menses
* HIV-1 seronegative at screening
* Normal Pap smear at screening or documented normal Pap smear within six months prior to screening
* No evidence of reproductive tract infection (RTI)
* Willing and able to comply with study procedures, including pelvic exams, colposcopy, maintaining a study coital and symptom log, and applying assigned study gel per protocol
* Agree to abstain from sexual intercourse for 24 hours prior to the enrollment visit
* Agree to abstain from the following activities from at least 48 hours prior to enrollment through the Day 14 visit:

  * Insertion of fingers and other objects into the vagina
  * Receiving oral sex
  * Receiving anal sex
  * Using a diaphragm, cervical cap, female condom, or vaginal contraceptive ring
  * Using vaginal products other than the study gels, including douches, lubricants, or feminine hygiene products
* In a monogamous sexually active relationship with one male partner
* Report having vaginal intercourse only with that partner at least two times per week
* No other reported partner in the prior six months and no plan to have another partner for the duration of the study
* Agree to use condoms for each act of vaginal intercourse during participation in the study
* Their male partner is informed and also consents to participate in the study
* Willing to have male partner informed and treated if an STD is diagnosed at screening or during the study

Inclusion Criteria for men:

* Age 18 years or older
* HIV-seronegative and free of other STI at screening exam
* One female sexual partner; no other reported partner in the prior six months and no plan to have another partner for the duration of the study
* Willing and able to comply with study procedures, including clinic visits, interviews and acceptability evaluation, and consistent use of condoms during enrollment in the study
* Willing to have female partner informed and treated if an STD is diagnosed at screening or during the study

Exclusion Criteria for women:

* Pregnancy or desire to become pregnant at time of study participation
* Currently breastfeeding
* Delivery or abortion within last eight weeks
* History of any male sexual partner other than current partner in past six months

  - No abnormal (DAIDS grade 1 or higher) laboratory results at baseline, including hematology, liver and kidney function
* History of post-coital vaginal bleeding in the past three months
* History of surgery to remove uterus or cervix
* History of surgery on the external genitalia, vaginal, or cervix in the past month
* Clinically significant chronic medical condition that is considered progressive, including cardiopulmonary disease, renal disease, hepatic disease, diabetes mellitus.
* History of sensitivity/allergy to latex
* Existence of a clinically detectable genital abnormality at screening (e.g. ulcer, congenital abnormality, any lesion with mucosal disruption)
* Concurrent participation in another trial of a vaginal product
* Have any other condition that in the opinion of the investigator might interfere with the evaluation of the study objectives

Exclusion Criteria for men:

* History of genital surgery in the past month
* Clinical or laboratory evidence of an STI.
* History of sensitivity/allergy to latex
* History of any sexual partner other than their current partner in the past six months

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2007-06; Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
Genital tract inflammation or epithelial disruption as assessed by naked eye and colposcopic inspection according to established guidelines | 2 weeks
Symptoms of irritation | two weeks
Changes in vaginal flora | Two weeks
Assessment of pro-inflammatory cytokines in the genital tract | Two weeks
Other product-related adverse events | Two weeks

SECONDARY OUTCOMES:
acceptability of UC-781 gel use | Two weeks
systemic absorption of UC-781 | Two weeks
anti-HIV activity of genital secretions in the presence of UC-781 gel | Two weeks

CONTACTS AND LOCATIONS:
Overall Officials: Sara J Whitehead, MD, MPH, Principal Investigator — Centers for Disease Control and Prevention; Chitlada Utaipiboon, MD, Principal Investigator — Thailand MOPH - U.S. CDC Collaboration
Locations (1):
- Chiang Rai Health Club, Chiang Rai, Thailand